CLINICAL TRIAL: NCT04927013
Title: Testing a Low Cost Population- and Theory-Based Outreach Intervention to Engage Ovarian Cancer Survivors and Their Close Relatives to Consider Genetic Services
Brief Title: Connecting Families to Overcome Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yue Guan, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00000224; 1U01CA240581 (NIH)
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Ovarian Cancer
Keywords: Genetic counseling; Risk assessment; Family communication; Genetic risk communication
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Message-based Outreach Intervention (MBI) for Survivors (Experimental): Cancer survivors randomized to receive a targeted letter with a unique website login code, access to the expanded website, free genetic counseling, and short message service (SMS) reminders.
  Interventions: Behavioral: Message-based Outreach Intervention for Survivors
- Standard Outreach for Survivors (Active Comparator): Cancer survivors randomized to receive the standard outreach consisting of a standard letter with website access, access to a condensed version of the study website, and free genetic counseling.
  Interventions: Behavioral: Standard Outreach for Survivors
- Message-based Outreach Intervention for Close Relatives (Experimental): Close relatives of cancer survivors who were randomized to receive the message-based outreach. Close relatives will have access to the expanded version of the study website and free genetic counseling.
  Interventions: Behavioral: Message-based Outreach Intervention for Close Relatives
- Standard Outreach for Close Relatives (Active Comparator): Close relatives of cancer survivors who were randomized to receive the standard outreach. Close relatives will have access to a condensed version of the study website and free genetic counseling.
  Interventions: Behavioral: Standard Outreach for Close Relatives

INTERVENTIONS:
Behavioral: Message-based Outreach Intervention for Survivors — The Georgia Cancer Registry will mail the initial recruitment containing messages intended to persuade the survivor to visit the study website as well as a unique login to access the website. In addition to the components of the standard website, an expanded website for the Message-based group will include Guidance for Talking with Close Relatives about Their Cancer Risk, and the request to enumerate each close relative and choose from a menu of options about how the survivor would prefer for their relatives to be contacted. Survivors also can select the option that they prefer a relative not be contacted. In this case, no invitation letter will be generated for these relatives. Survivors who provide mobile phone numbers will receive two SMS thanking them for accessing the website, and encouraging them to revisit the website to review information and contact relatives. The messages will occur at 3-week intervals over a 6-week time period.
  Arms: Message-based Outreach Intervention (MBI) for Survivors
Behavioral: Standard Outreach for Survivors — The Georgia Cancer Registry will mail survivors an introductory letter modeled on the Registry's general outreach letters that will include log in information. Survivors will have access to a condensed version of the website that includes Information about Ovarian Cancer, Information about Who in Your Family is at Increased Risk, and the offer of Free Genetic Counseling with the option to schedule an appointment.
  Arms: Standard Outreach for Survivors
Behavioral: Message-based Outreach Intervention for Close Relatives — Relatives will receive a unique website login linked to the survivor that enables access to the website. The website content will be identical to the survivor content with the exception of the addition of the Breast Cancer Genetics Referral Screening Tool (B-RST) risk assessment tool. This brief risk assessment is a validated screening tools that is clinically useful for estimating the probability of breast cancer (BRCA1/2) gene mutation and identifying women for referral to genetic counseling. Although all 1st or 2nd degree relatives of ovarian cancer survivors will screen positive on B-RST, asking relatives to complete the screener aims to raise their awareness of the factors that contribute to hereditary risk of ovarian cancer and will reinforce the salience of seeking genetic counseling. Additionally, relatives for who provide cell phone numbers will receive 3 SMS reminders over 9 weeks.
  Arms: Message-based Outreach Intervention for Close Relatives
Behavioral: Standard Outreach for Close Relatives — The invitation letter shared by the survivor will provide a unique login code for each relative to visit the standard website with sections specifically for relatives that include information about genetic risk, the value of completing an online short validated risk screener, and the offer of free genetic counseling with the option to schedule an appointment.
  Arms: Standard Outreach for Close Relatives

SUMMARY:
This study tests a multi-component, low cost, message-based communication outreach intervention to engage ovarian cancer survivors and their at-risk relatives in considering cancer genetic services. The intervention includes foot-in-the-door techniques, tailored/targeted print, website support, and short messages to expand reach of prevention messages.

DETAILED DESCRIPTION:
The majority of women at greatest risk for ovarian cancer due to hereditary factors are unlikely to be aware of their elevated risk and available prevention options. Thus, most at-risk women are diagnosed when their ovarian cancer is advanced and treatment options are limited. Additionally, efforts to broaden awareness of genetic risk among at risk families has been very limited. State cancer registries' offer a potentially low cost platform for providing resources to ovarian cancer survivors and their close relatives.

In partnership with the Georgia Cancer Registry (GCR), the researchers are testing two different communication approaches to provide inherited risk information and free genetic counseling to ovarian cancer survivors and their close blood relatives. Participants will be assigned at random to visit one of two websites; those assigned to the "message-based" site will be offered assistance from the study team to contact close relatives and reminder messages and those viewing the other site will not. The researchers are testing which of the two approaches is most effective as indicated by: the number of survivors who visit the website; the number of close relatives who visit the website and the number of survivors and relatives who complete a genetic counseling session. The researchers hypothesize that the message-based approach will result in greater reach and uptake of genetic services than a standard approach.

The two outreach websites with content for both survivors and close relatives will be the hub in the wheel of intervention activity. In turn, the researchers will encourage access to the website using other communication channels as the spokes. The GCR will make initial contact with ovarian cancer survivors. The Registry will: 1) mail a packet of information about the study to identified survivors, and 2) make follow-up phone calls and send reminder postcards to encourage study participation. Survivors can then visit the assigned website and click a button indicating they agree to participate. Survivors assigned to the message-based intervention will receive additional short text messages encouraging them to contact relatives and seek genetic counseling. Relatives in this message-based group who choose to participate will also receive these short messages if they choose to provide contact information.

Free genetic counseling is being offered to participants in both study arms. The researchers are collaborating with Emory's Genetic Counseling Training program under the supervision of two certified genetic counselors. This study uses tele-medicine approaches to ensure access of survivors and relatives living in Georgia and elsewhere.

The results of the study could guide the development of outreach strategies for Georgia and other states to offer sustainable services to expand the reach of genetic services for ovarian and other heritable cancers.

ELIGIBILITY:
Inclusion Criteria for Survivors:

* in the Georgia Cancer Registry (GSR)
* diagnosed with ovarian, fallopian tube, or peritoneal cancers
* lived in Georgia at the time of diagnosis
* not deceased per the registry's records
* have a mailing address in GSR records

Inclusion Criteria for Close Relatives:

* 25 years or older
* able to access the internet
* a 1st or 2nd degree relative of the survivor
* able to read English
* non-incarcerated or institutionalized

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2331 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McBride, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available for sharing, after de-identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for sharing immediately following the publication and release of the key manuscripts tied to the primary aims of this study, and ending approximately 18 months after funding ends.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims stated in the approved proposal. Proposals should be directed to Dr. Colleen McBride at colleen.marie.mcbride@emory.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Guan Y, McBride CM, Zhao J, Pentz RD, Escoffery C, Liu Y, Cao Y, An W, Shepperd JA, Ward KC. Testing a Population-Based Outreach Intervention for Ovarian Cancer Survivors to Encourage their Close Relatives to Consider Genetic Counseling. Cancer Epidemiol Biomarkers Prev. 2024 Sep 3;33(9):1185-1193. doi: 10.1158/1055-9965.EPI-24-0147. PMID 38912902
- [Derived] Shepperd JA, McBride CM, An W, Zhao J, Pentz RD, Escoffery C, Ward K, Guan Y. Trust and Privacy Concerns Among Cancer Survivors Who Did Not Visit a Research Website Offering Free Genetic Counseling Services for Families: Survey Study. J Med Internet Res. 2025 May 6;27:e64228. doi: 10.2196/64228. PMID 40327861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began July 24, 2021 and all follow up was complete by February 21, 2023. Participants were identified from the Georgia Cancer Registry (GCR) which includes persons diagnosed with cancer in the state of Georgia, USA.
Groups:
- Message-based Outreach Intervention (MBI) for Survivors: Cancer survivors randomized to receive a targeted letter with a unique website login code, access to the expanded website, free genetic counseling, and short message service (SMS) reminders.
  Message-based Outreach Intervention for Survivors: The Georgia Cancer Registry will mail the initial recruitment containing messages intended to persuade the survivor to visit the study website as well as a unique login code to access the website. In addition to the components of the standard website, an expanded website for the Message-based group will include Guidance for Talking with Close Relatives about Their Cancer Risk, and the request to enumerate each close relative and choose from a menu of options about how the survivor would prefer for their relatives to be contacted. Survivors also can select the option that they prefer a relative not be contacted. In this case, no invitation letter will be generated for these relatives. Survivors who provide mobile phone numbers will receive two SMS thanking them for accessing the website, and encouraging them to revisit the website to review information and contact relatives. The messages will occur at 3-week intervals over a 6-week time period.
- Standard Outreach for Survivors: Cancer survivors randomized to receive the standard outreach consisting of a standard letter with a unique website login code, access to a condensed version of the study website, and free genetic counseling.
  Standard Outreach for Survivors: The Georgia Cancer Registry will mail survivors an introductory letter modeled on the Registry's general outreach letters that will include log in information. Survivors will have access to a condensed version of the website that includes Information about Ovarian Cancer, Information about Who in Your Family is at Increased Risk, and the offer of Free Genetic Counseling with the option to schedule an appointment.
- Message-based Outreach Intervention for Close Relatives: Close relatives of cancer survivors who were randomized to receive the message-based outreach. Close relatives will have access to the expanded version of the study website and free genetic counseling.
  Message-based Outreach Intervention for Close Relatives: Relatives will receive a unique website login code linked to the survivor that enables access to the website. The website content will be identical to the survivor content with the exception of the addition of the Breast Cancer Genetics Referral Screening Tool (B-RST) risk assessment tool. This brief risk assessment is a validated screening tools that is clinically useful for estimating the probability of breast cancer (BRCA1/2) gene mutation and identifying women for referral to genetic counseling. Although all 1st or 2nd degree relatives of ovarian cancer survivors will screen positive on B-RST, asking relatives to complete the screener aims to raise their awareness of the factors that contribute to hereditary risk of ovarian cancer and will reinforce the salience of seeking genetic counseling. Additionally, relatives for who provide cell phone numbers will receive 3 SMS reminders over 9 weeks.
- Standard Outreach for Close Relatives: Close relatives of cancer survivors who were randomized to receive the standard outreach. Close relatives will receive a unique login code to access a condensed version of the study website and free genetic counseling.
  Standard Outreach for Close Relatives: The invitation letter shared by the survivor will provide a unique login code for each relative to visit the standard website with sections specifically for relatives that include information about genetic risk, the value of completing an online short validated risk screener, and the offer of free genetic counseling with the option to schedule an appointment.
Period: Overall Study
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives
Started (Cancer survivors considered as starting the study are individuals from the GCR who were randomized to a study arm. Close relatives who started the study are individuals who were identified by survivors who used their unique login code to access the study website.) | 969 | 969 | 152 | 241
Completed (Individuals who started the study are considered as completing the study if they consented to participate while they were using the website.) | 130 | 184 | 19 | 1
Not Completed | 839 | 785 | 133 | 240

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes cancer survivors who gave consent to participate in the study. Baseline characteristics were not collected for close relatives.
Groups:
- Standard Outreach for Survivors: Cancer survivors randomized to receive the standard outreach consisting of a standard letter with a unique website login code, access to a condensed version of the study website, and free genetic counseling.
- Total: Total of all reporting groups
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives | Total
Number analyzed (Participants) | 130 | 184 | 0 | 0 | 314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 73 | 93 |  |  | 166
  >=65 years | 57 | 91 |  |  | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (13.0) | 63.5 (12.5) |  |  | 63.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 184 |  |  | 314
  Male | 0 | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 |  |  | 9
  Not Hispanic or Latino | 126 | 179 |  |  | 305
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 1 | 3 |  |  | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 28 | 32 |  |  | 60
  White | 101 | 149 |  |  | 250
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130 | 184 |  |  | 314
Age at diagnosis [Mean (Standard Deviation); unit: years] | 52.7 (12.6) | 53.6 (12.6) |  |  | 53.3 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Survivors Using Website Access Code
Description: Survivor reach is assessed as the number of the eligible survivors identified and contacted by GCR who used their unique login to access the study website.
Time Frame: Up to 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors
Number analyzed (Participants) | 969 | 969
Participants | 147 | 202

2. Primary Outcome: Number of Survivors Consenting to Participate in the Study
Description: Survivor reach is assessed as the number of the eligible survivors identified and contacted by GCR who used their unique login code to access the study website and consented to participate in the study while visiting the website.
Time Frame: Up to 19 months
Population: The analysis population includes individuals who used their unique login code to access the study website.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors
Number analyzed (Participants) | 147 | 202
Participants | 130 | 184

3. Primary Outcome: Number of Survivors Creating a Study Login
Description: Survivor reach is assessed as the number of the eligible survivors identified and contacted by GCR who access the study website, consented to participate in the study, and created their own personal study login on the website.
Time Frame: Up to 19 months
Population: The analysis population includes individuals who gave consent to participate in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors
Number analyzed (Participants) | 130 | 184
Participants | 126 | 174

4. Primary Outcome: Number of Relatives of Survivors Using the Website Access Code
Description: Close relative reach is assessed as the number of close relatives enumerated by survivors who used their unique login code to access the study website.
Time Frame: Up to 19 months
Population: The analysis population includes close relatives of cancer survivors who were identified by the survivors to be contacted and offered the opportunity to participate in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives
Number analyzed (Participants) | 152 | 241
Participants | 20 | 1

5. Primary Outcome: Number of Relatives of Survivors Consenting to Participate in the Study
Description: Close relative reach is assessed as the number of close relatives enumerated by survivors who accessed the website and consented to participate in the study while they were using the website.
Time Frame: Up to 19 months
Population: The analysis population includes close relatives who accessed the study website.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives
Number analyzed (Participants) | 20 | 1
Participants | 19 | 1

6. Primary Outcome: Number of Relatives of Survivors Creating a Login
Description: Close relative reach is assessed as the number of close relatives enumerated by survivors who accessed the study website, gave consent to participate in the study, and created their own personal study login on the study website.
Time Frame: Up to 19 months
Population: This analysis population includes close relatives who gave consent to participate in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives
Number analyzed (Participants) | 19 | 1
Participants | 19 | 0

7. Secondary Outcome: Relative Contact Option Selected by Survivors
Description: Cancer survivors in the Message-based Outreach Intervention arm who accessed the website were asked to enumerate close relatives and choose from a menu of options about how the survivor would prefer for their relatives to be contacted.
Time Frame: Up to 19 months
Population: This analysis population includes cancer survivors who accessed the website and selected a contact method for the close relatives that they provided contact information for. Survivors could identify more than one close relative and some did not identify any relatives.
Measure: Count of Participants; unit: Participants
Groups:
- Message-based Outreach Intervention for Survivors: Cancer survivors randomized to receive a targeted letter with a unique website login code, access to the expanded website, free genetic counseling, and short message service (SMS) reminders.
Arm/Group | Message-based Outreach Intervention for Survivors
Number analyzed (Participants) | 136
Participants
  Survivor Participant Selected "Self-Contact" | 78
  Survivor Participant Selected "Study Team Contact" | 34
  Survivor Participant Selected "Delay Contact" | 24

8. Secondary Outcome: Number of Survivors Requesting Telegenetic Counseling
Description: The request rate of cancer genetic services is assessed as the number of cancer survivors who requested telegenetic counseling on the website.
Time Frame: Up to 19 months
Population: This analysis includes participants who accessed the study website.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors
Number analyzed (Participants) | 147 | 202
Participants | 26 | 17

9. Secondary Outcome: Number of Survivors Completing Telegenetic Counseling
Description: Uptake of cancer genetic services is assessed as the number of survivors who completed telegenetic counseling.
Time Frame: Up to 19 months
Population: This analysis includes participants who requested telegenetic counseling on the website.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors
Number analyzed (Participants) | 26 | 17
Participants | 15 | 9

10. Secondary Outcome: Number of Relatives Requesting Telegenetic Counseling
Description: The request rate of cancer genetic services is assessed as the number of close relatives who requested telegenetic counseling on the website.
Time Frame: Up to 19 months
Population: This analysis population includes close relatives who gave consent to participate in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives
Number analyzed (Participants) | 19 | 1
Participants | 9 | 0

11. Secondary Outcome: Number of Relatives Completing Telegenetic Counseling
Description: Uptake of cancer genetic services by relatives of survivors is assessed as the number of relatives enumerated who completed the Breast Cancer Genetics Referral Screening Tool (B-RST) screening and subsequently accessed genetic counseling.
Time Frame: Up to 19 months
Population: This analysis includes relatives who requested telegenetic counseling on the website.
Measure: Count of Participants; unit: Participants
Arm/Group | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives
Number analyzed (Participants) | 9 | 0
Participants | 8 | 0

12. Secondary Outcome: Time Visiting Website by Survivors
Description: The duration of time (in minutes) that survivors in the Message-based Outreach Intervention (MBI) study arm spent on the website was examined.
Time Frame: Up to 19 months
Population: The analysis population includes survivors in the MBI study arm who created a personal study login and used the website. Ten participants had no website activity after creating their login.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors
Number analyzed (Participants) | 116
minutes | 14.81 (15.68)

13. Secondary Outcome: Time Visiting Website by Relatives
Description: Among those in the intervention arm, the duration of time (in minutes) that relatives of survivors spend on the website was examined.
Time Frame: Up to 19 months
Population: The analysis population includes close relatives of survivors in the MBI study arm who gave consent to participate in the study.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Message-based Outreach Intervention for Close Relatives
Number analyzed (Participants) | 19
minutes | 6.78 (3.42)

14. Secondary Outcome: Number of Return Visits to Website by Survivors
Description: The number of return visits to the website by survivors in the MBI study arm was examined.
Time Frame: Up to 19 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: return visits
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors
Number analyzed (Participants) | 116
return visits | 1.56 (1.25)

15. Secondary Outcome: Number of Return Visits to Website by Relatives
Description: Among those in the intervention arm, the number of return visits to the website by relatives of survivors was examined.
Time Frame: Up to 19 months
Population: This analysis population includes close relatives of survivors in the MBI study arm who gave consent to participate in the study.
Measure: Mean (Standard Deviation); unit: return visits
Arm/Group | Message-based Outreach Intervention for Close Relatives
Number analyzed (Participants) | 19
return visits | 1.31 (0.58)

16. Secondary Outcome: Number of Pages Viewed by Survivors
Description: The number of website page viewed by survivors in the MBI study arm was examined.
Time Frame: Up to 19 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: number of pages viewed
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors
Number analyzed (Participants) | 116
number of pages viewed | 10.25 (7.99)

17. Secondary Outcome: Number of Pages Viewed by Relatives
Description: Among those in the intervention arm, the number of website pages viewed by relatives of survivors will be examined.
Time Frame: Up to 19 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: number of pages viewed
Arm/Group | Message-based Outreach Intervention for Close Relatives
Number analyzed (Participants) | 19
number of pages viewed | 13.37 (3.83)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning when the study intervention began through the final study assessment (up to 19 months).
Arm/Group | Message-based Outreach Intervention (MBI) for Survivors | Standard Outreach for Survivors | Message-based Outreach Intervention for Close Relatives | Standard Outreach for Close Relatives
All-Cause Mortality (participants affected / at risk) | 0/969 | 0/969 | 0/152 | 0/241
Serious Adverse Events (participants affected / at risk) | 0/969 | 0/969 | 0/152 | 0/241
Other Adverse Events (participants affected / at risk) | 0/969 | 0/969 | 0/152 | 0/241

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT04927013/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT04927013/ICF_000.pdf